CLINICAL TRIAL: NCT00726726
Title: Effect of Concomitant Administration of BMS-708163 on the Pharmacokinetics of Midazolam, Warfarin, Caffeine, Omeprazole and Dextromethorphan in Healthy Male Subjects by Administration of a Modified Cooperstown Cocktail
Brief Title: Drug Interaction Study With a Potential Alzheimer's Disease Compound
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN156-005
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2008-11-05 (Estimated); Status verified 2008-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Midazolam; Warfarin; Vitamin K; Caffeine; Omeprazole; Dextromethorphan; BMS 708163

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Other)
  Interventions: Drug: Interacting drugs - Cooperstown Cocktail (midazolam, warfarin, (+ vitamin K), caffeine, omeprazole and dextromethorphan)
- B (Experimental)
  Interventions: Drug: BMS-708163
- C (Experimental): + Other
  Interventions: Drug: BMS-708163 + Cooperstown Cocktail

INTERVENTIONS:
Drug: Interacting drugs - Cooperstown Cocktail (midazolam, warfarin, (+ vitamin K), caffeine, omeprazole and dextromethorphan) — Capsules + Tablets + Oral solution, Oral, Midazolam: 5 mg, Warfarin: 10 mg (vitamin K 10 mg), caffeine: 200 mg, omeprazole: 40 mg, dextromethorphan: 30 mg once daily, Day 1, 1 Day
  Arms: A
Drug: BMS-708163 — Capsules, Oral, 150 mg, once daily, days 6-15, 10 Days
  Arms: B
Drug: BMS-708163 + Cooperstown Cocktail — Capsules + tablets + Oral solution, Oral, BMS-708163: 150 mg + Midazolam: 5 mg, Warfarin: 10 mg (vitamin K 10 mg), caffeine: 200 mg, omeprazole: 40 mg, dextromethorphan: 30 mg, BMS-708163, once daily, days 16-20 midazolam,warfarin, (+ vitamin K), caffeine, omeprazole and dextromethorphan once daily on Day 16, 5 Days
  Arms: C

SUMMARY:
The purpose of this study is to determine whether BMS-708163 will effect the pharmacokinetics of the commonly prescribed medicines midazolam, warfarin, caffeine,omeprazole and dextromethorphan

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* 18-45 yrs old inclusive

Exclusion Criteria:

* Women

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic effects of BMS-708163 on interacting drugs (midazolam, warfarin, caffeine, omeprazole, and dextromethorphan) | throughout the study

SECONDARY OUTCOMES:
Safety variables (adverse events, vital signs, safety labs) | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bristol-Myers Squibb Clinical Pharmacology Unit, Hamilton, New Jersey, United States